CLINICAL TRIAL: NCT07302971
Title: Telemedicine-supported Management of Acute Ischemic Stroke in the Basic-level Hospitals
Brief Title: Telemedicine-supported Management for Acute Ischemic Stroke
Acronym: TOGETHER
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Capital Medical University (Other)
Responsible Party: Principal Investigator, Ji Xunming,MD,PhD, Professor of Neurology, Xuanwu Hospital, Capital Medical University, Capital Medical University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: TOGETHER
Record Dates: First submitted 2025-12-02; First posted 2025-12-24 (Actual); Last update posted 2026-02-03 (Actual); Status verified 2025-11

CONDITIONS: Acute Ischemic Stroke
MeSH Terms: conditions — Ischemic Stroke

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Telemedicine-Supported Group (Experimental): Receive remote guidance from expert stroke centers for treatment of patients with intravenous thrombolysis, along with quality control for standardized workflow support, and professional training.
  Interventions: Other: Telemedicine-Supported Management
- Standard Treatment Group without Telemedicine-Supported Management (No Intervention): Control-group patients will receive routine stroke care at their primary care hospitals, with no remote consultation, study-related quality control, or extra training. Care will follow the hospitals' usual protocols, including emergency assessment, neurological evaluation, imaging, and intravenous thrombolysis. Hospitals may continue their regular stroke-related training during the study to reflect real-world practice.

INTERVENTIONS:
Other: Telemedicine-Supported Management — Receive round-the-clock 7×24h remote consultation guidance from expert teams at leading stroke centers, covering patient triage and initial assessment, thrombolysis decision-making, and treatment guidance. Undergo quality control for standardized workflow implementation, and professional training.
  Arms: Telemedicine-Supported Group

SUMMARY:
Telemedicine-supported stroke care can provide standardized guidance to hospitals and regions with limited medical resources, thereby improving treatment outcomes for stroke patients in these areas. While this approach has been widely adopted in many developed countries, its efficacy in guiding basic-level hospitals to manage acute ischemic stroke requires further investigation through large-scale, high-quality studies.

This study focused on patients with acute ischemic stroke who sought treatment at basic-level hospitals, aiming to investigate the efficacy and safety of treating acute ischemic stroke with telemedicine-supported management. Hospitals assigned to the experimental group received remote consultation guidance, quality control and professional training from expert teams at leading stroke centers, China National Center for Neurological Disorders. Hospitals in the control group did not receive telemedicine-supported management.

ELIGIBILITY:
Inclusion Criteria:

* Hospital Inclusion Criteria:

  1. Basic-level hospitals in China (Definition: Hospitals classified as secondary-level (Grade II) or below under China's Hospital Grading Management Standards, or hospitals located in counties/county-level cities).
  2. Equipped with an emergency department and neurology ward capable of admitting stroke patients.
  3. Equipped with CT and/or MRI capable of diagnosing AIS.
  4. Equipped with intravenous thrombolytic drugs for acute ischemic stroke.
* Patient Inclusion Criteria:

  1. Age ≥ 18 years.
  2. Diagnosed with acute ischemic stroke.
  3. CT/MRI confirms absence of intracerebral hemorrhage.
  4. Onset of stroke symptoms ≤ 4.5 hours.
  5. pre-stroke mRS score ≤1.
  6. Informed consent obtained from patient or their legal representative.

Exclusion Criteria:

* Hospital Exclusion Criteria:

  1. Admitting fewer than 10 patients with acute ischemic stroke per month.
  2. Currently participating in other clinical trials that may interfere with this trial.
* Patient Exclusion Criteria:

  1. Presence of contraindications for intravenous thrombolysis according to AHA/ASA guidelines

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2400 (Estimated)
Dates: Start 2026-02-02 (Actual); Primary Completion 2027-06 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Proportion of patients with mRS scores of 0-1 | 90 days

SECONDARY OUTCOMES:
Intravenous thrombolysis rate | 4.5 hours
mRS score | 90 days
  Ranges from 0 to 6 points, with lower scores indicating better functional outcome.
Door-to-(thrombolysis)needle-time | 4.5 hours
  The time calculation begins when the patient arrives at the hospital and ends upon receiving thrombolytic therapy. The theoretical range is 0 to 270 minutes.
Rate of endovascular therapy receipt among eligible patients | 24 hours

OTHER OUTCOMES:
Proportion of sICH | Within 36 hours of thrombolysis
  The time frame is within 36 hours after thrombolysis in patients. Symptomatic intracranial hemorrhage occurring during this period is considered an endpoint event. If the patient is discharged within 36 hours, the endpoint event is observed during the hospitalization period.
Proportion of any type of ICH | Within 36 hours of thrombolysis
  The time frame is within 36 hours of thrombolysis administration. Any type of intracerebral hemorrhage occurring during this period is considered an endpoint event. If the patient is discharged within 36 hours, the endpoint event is observed during the hospitalization period.
All-cause mortality rate | 90 days

CONTACTS AND LOCATIONS:
Locations (1):
- Xuanwu Hospital, Beijing, Beijing Municipality, China